CLINICAL TRIAL: NCT06061653
Title: Effects of Augmentation of Interpersonal Psychotherapy With High-Definition Transcranial Direct Current Stimulation for Adolescent Depression: A Randomized Clinical Trial
Brief Title: Augmentation of Interpersonal Psychotherapy With High-Definition Transcranial Direct Current Stimulation for Adolescent Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIT2023496
Record Dates: First submitted 2023-08-08; First posted 2023-09-29 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-05

CONDITIONS: Depressive Disorder
MeSH Terms: conditions — Depressive Disorder | interventions — adenylate isopentenyltransferase

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPT plus HD-tDCS (Experimental)
  Interventions: Combination Product: IPT plus HD-tDCS
- IPT plus sham HD-tDCS (Sham Comparator)
  Interventions: Combination Product: IPT plus sham HD-tDCS

INTERVENTIONS:
Combination Product: IPT plus HD-tDCS — psychotherapy plus device
  Arms: IPT plus HD-tDCS
Combination Product: IPT plus sham HD-tDCS — psychotherapy plus sham device
  Arms: IPT plus sham HD-tDCS

SUMMARY:
Depression is among the most prevalent psychiatric disorders, with an upward trend in its manifestation in younger individuals. In contrast to adult depression, adolescent depression often presents with longer attack durations, higher recurrence rates, chronicity, and elevated disability rates. At present, treatment options for adolescent depression encompass pharmacological, physical, and psychological therapies. However, current evidence suggests that no antidepressant medication is entirely safe for youths, with only fluoxetine and escitalopram being FDA-approved for treating adolescent depression.

Given the weight of interpersonal stressors faced by teenagers, the NICE guidelines recommend interpersonal therapy(IPT) as a first-line treatment. A 2020 meta-analysis in the Journal of the American Academy of Child and Adolescent Psychiatry reported that interpersonal therapy exhibited significantly greater improvements in depression symptoms than cognitive behavioral therapy(CBT), although psychotherapeutic effects were modest, achieving a remission rate of 60%. These results underscore the need for further research to enhance interpersonal therapy's effectiveness in treating adolescent depression.

High-Definition Transcranial Direct Current Stimulation (HD-tDCS）is a highly secure non-invasive brain stimulation technique that produces sustained effects even after stimulation has discontinued, rendering it particularly valuable for therapeutic interventions. The proposed study aims to augment a single IPT treatment with HD-tDCS stimulation for adolescent depression. By enhancing the excitability of the cerebral cortex, HD-tDCS could potentially enhance IPT's therapeutic efficacy in treating adolescent depression while facilitating further investigation of its underlying neural circuit mechanisms.

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent form, willing to participate in the study and accept treatment (patients under 18 years of age need to obtain the consent of their parents or legal guardians);
2. Age between 12 and 18 years;
3. Right-handed;
4. Han ethnicity;
5. Meet the DSM-5 diagnostic criteria for depression;
6. HAMD-24≥20;
7. Understand written language and able to complete questionnaires;
8. First-episode depression patients who have never received any treatment or relapse depression patients, have not taken any psychotropic drugs in the past 2 weeks, have not received systematic psychological or physical therapy.

Exclusion Criteria:

1. Exclusion criteria for tDCS: (1) Patients with metal implants in the body; those with metal implants such as titanium or magnetic devices (including aneurysm clips); (2) Patients with implanted devices such as cardiac pacemakers, deep brain stimulators (DBS); (3) Patients with intracranial hypertension, skull defects, or tumors; (4) Patients with unstable vital signs such as severe cardiac or somatic diseases; (5) Patients in the acute phase of cerebrovascular diseases; (6) Patients with adverse reactions to electrical stimulation; (7) Patients with pain sensitivity, injury, or inflammation in the stimulation area.
2. Exclusion criteria for MRI;
3. Patients with severe neurological, cardiac, liver, kidney, endocrine, and blood system diseases, or any other condition that may interfere with the study evaluation;
4. Patients with organic mental disorders and mental retardation;
5. Patients with alcohol or drug dependence;
6. Patients with a high risk of suicide.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
24-item Hamilton Depression Rating Scale | Baseline
  Assessment of depressive symptoms. Score<8: normal; >20: mild or moderate depression; >35: severe depression.
24-item Hamilton Depression Rating Scale | 1-month
  Assessment of depressive symptoms. Score<8: normal; >20: mild or moderate depression; >35: severe depression.
24-item Hamilton Depression Rating Scale | 2-month
  Assessment of depressive symptoms. Score<8: normal; >20: mild or moderate depression; >35: severe depression.
24-item Hamilton Depression Rating Scale | 3-month
  Assessment of depressive symptoms. Score<8: normal; >20: mild or moderate depression; >35: severe depression.
Child Depression Rating Scale-Revised | Baseline
  Assessment of depressive symptoms. Score<40: normal; 40~60: mild or moderate depression; >60: severe depression.
Child Depression Rating Scale-Revised | 1-month
  Assessment of depressive symptoms. Score<40: normal; 40~60: mild or moderate depression; >60: severe depression.
Child Depression Rating Scale-Revised | 2-month
  Assessment of depressive symptoms. Score<40: normal; 40~60: mild or moderate depression; >60: severe depression.
Child Depression Rating Scale-Revised | 3-month
  Assessment of depressive symptoms. Score<40: normal; 40~60: mild or moderate depression; >60: severe depression.

SECONDARY OUTCOMES:
17-item Hamilton Anxiety Rating Scale | Baseline
  Score<7:No anxiety; Score≥7:Possibly anxious; Score≥14:Definitely anxious; Score≥21:Definitely significantly anxious; Score≥29:Possibly severely anxious.
17-item Hamilton Anxiety Rating Scale | 1-month
  Score<7:No anxiety; Score≥7:Possibly anxious; Score≥14:Definitely anxious; Score≥21:Definitely significantly anxious; Score≥29:Possibly severely anxious.
17-item Hamilton Anxiety Rating Scale | 2-month
  Score<7:No anxiety; Score≥7:Possibly anxious; Score≥14:Definitely anxious; Score≥21:Definitely significantly anxious; Score≥29:Possibly severely anxious.
17-item Hamilton Anxiety Rating Scale | 3-month
  Score<7:No anxiety; Score≥7:Possibly anxious; Score≥14:Definitely anxious; Score≥21:Definitely significantly anxious; Score≥29:Possibly severely anxious.
Beck Scale for Suicide Ideation | Baseline
  Assessment of suicidal ideation. The test taker first completes the initial five questions. If the responses to both the fourth and fifth items are "no," it is considered that there is no suicidal ideation, and the questionnaire concludes. Suicidal risk is evaluated based on items six to nineteen of the scale, which assess the likelihood of actual suicidal behavior among individuals with suicidal ideation. The calculation formula for the total score is [(sum of scores for items six to nineteen) - 9) / 33] * 100, resulting in a score ranging from 0 to 100. A higher score indicates a greater risk of suicide.
Beck Scale for Suicide Ideation | 1-month
  Assessment of suicidal ideation. The test taker first completes the initial five questions. If the responses to both the fourth and fifth items are "no," it is considered that there is no suicidal ideation, and the questionnaire concludes. Suicidal risk is evaluated based on items six to nineteen of the scale, which assess the likelihood of actual suicidal behavior among individuals with suicidal ideation. The calculation formula for the total score is [(sum of scores for items six to nineteen) - 9) / 33] * 100, resulting in a score ranging from 0 to 100. A higher score indicates a greater risk of suicide.
Beck Scale for Suicide Ideation | 2-month
  Assessment of suicidal ideation. The test taker first completes the initial five questions. If the responses to both the fourth and fifth items are "no," it is considered that there is no suicidal ideation, and the questionnaire concludes. Suicidal risk is evaluated based on items six to nineteen of the scale, which assess the likelihood of actual suicidal behavior among individuals with suicidal ideation. The calculation formula for the total score is [(sum of scores for items six to nineteen) - 9) / 33] * 100, resulting in a score ranging from 0 to 100. A higher score indicates a greater risk of suicide.
Beck Scale for Suicide Ideation | 3-month
  Assessment of suicidal ideation. The test taker first completes the initial five questions. If the responses to both the fourth and fifth items are "no," it is considered that there is no suicidal ideation, and the questionnaire concludes. Suicidal risk is evaluated based on items six to nineteen of the scale, which assess the likelihood of actual suicidal behavior among individuals with suicidal ideation. The calculation formula for the total score is [(sum of scores for items six to nineteen) - 9) / 33] * 100, resulting in a score ranging from 0 to 100. A higher score indicates a greater risk of suicide.
the Chinese version of the Snaith-Hamilton Pleasure Scale | Baseline
  A total of 14 items, each with a score of 1 to 4, will be used to calculate the total score. The higher the score The higher the score, the more severe the pleasure deficit
the Chinese version of the Snaith-Hamilton Pleasure Scale | 1-month
  A total of 14 items, each with a score of 1 to 4, will be used to calculate the total score. The higher the score The higher the score, the more severe the pleasure deficit
the Chinese version of the Snaith-Hamilton Pleasure Scale | 2-month
  A total of 14 items, each with a score of 1 to 4, will be used to calculate the total score. The higher the score The higher the score, the more severe the pleasure deficit
the Chinese version of the Snaith-Hamilton Pleasure Scale | 3-month
  A total of 14 items, each with a score of 1 to 4, will be used to calculate the total score. The higher the score The higher the score, the more severe the pleasure deficit
Interpersonal Relationship Scale | Baseline
  A score of 0-8 indicates that interpersonal relationship is good, a score of 9-14 indicates that there is a certain degree of interpersonal relationship distress, and a score of 15-28 indicates that interpersonal relationship distress is more serious, that is, the lower the score of the comprehensive diagnostic scale of interpersonal relationship, the better the interpersonal relationship.
Interpersonal Relationship Scale | 1-month
  A score of 0-8 indicates that interpersonal relationship is good, a score of 9-14 indicates that there is a certain degree of interpersonal relationship distress, and a score of 15-28 indicates that interpersonal relationship distress is more serious, that is, the lower the score of the comprehensive diagnostic scale of interpersonal relationship, the better the interpersonal relationship.
Interpersonal Relationship Scale | 2-month
  A score of 0-8 indicates that interpersonal relationship is good, a score of 9-14 indicates that there is a certain degree of interpersonal relationship distress, and a score of 15-28 indicates that interpersonal relationship distress is more serious, that is, the lower the score of the comprehensive diagnostic scale of interpersonal relationship, the better the interpersonal relationship.
Interpersonal Relationship Scale | 3-month
  A score of 0-8 indicates that interpersonal relationship is good, a score of 9-14 indicates that there is a certain degree of interpersonal relationship distress, and a score of 15-28 indicates that interpersonal relationship distress is more serious, that is, the lower the score of the comprehensive diagnostic scale of interpersonal relationship, the better the interpersonal relationship.
Emotion Regulation Questionnaire | Baseline
  A total of 10 items were scored at 7 points. The higher the score, the higher the frequency of using emotion regulation strategies.
Emotion Regulation Questionnaire | 1-month
  A total of 10 items were scored at 7 points. The higher the score, the higher the frequency of using emotion regulation strategies.
Emotion Regulation Questionnaire | 2-month
  A total of 10 items were scored at 7 points. The higher the score, the higher the frequency of using emotion regulation strategies.
Emotion Regulation Questionnaire | 3-month
  A total of 10 items were scored at 7 points. The higher the score, the higher the frequency of using emotion regulation strategies.
Toronto Alexithymia Scale-20 | Baseline
  It consists of 3 factors, difficulty identifying feelings (DIF), difficulty describing feelings (DDF), and externally oriented thinking (EOT), which are called F1, F2, and F3 factors, containing 20 items, each scored within a 5-point scale (1: completely disagree to 5: completely agree), 20-100 points, the higher the score, the more pronounced the dysfunction in describing feelings.
Toronto Alexithymia Scale-20 | 1-month
  It consists of 3 factors, difficulty identifying feelings (DIF), difficulty describing feelings (DDF), and externally oriented thinking (EOT), which are called F1, F2, and F3 factors, containing 20 items, each scored within a 5-point scale (1: completely disagree to 5: completely agree), 20-100 points, the higher the score, the more pronounced the dysfunction in describing feelings.
Toronto Alexithymia Scale-20 | 2-month
  It consists of 3 factors, difficulty identifying feelings (DIF), difficulty describing feelings (DDF), and externally oriented thinking (EOT), which are called F1, F2, and F3 factors, containing 20 items, each scored within a 5-point scale (1: completely disagree to 5: completely agree), 20-100 points, the higher the score, the more pronounced the dysfunction in describing feelings.
Toronto Alexithymia Scale-20 | 3-month
  It consists of 3 factors, difficulty identifying feelings (DIF), difficulty describing feelings (DDF), and externally oriented thinking (EOT), which are called F1, F2, and F3 factors, containing 20 items, each scored within a 5-point scale (1: completely disagree to 5: completely agree), 20-100 points, the higher the score, the more pronounced the dysfunction in describing feelings.
The Reflective Function Questionnaire for Youths | Baseline
  Assesses the degree of agreement or disagreement with narratives about reflective functioning, with higher scores representing higher levels of reflective functioning.
The Reflective Function Questionnaire for Youths | 1-month
  Assesses the degree of agreement or disagreement with narratives about reflective functioning, with higher scores representing higher levels of reflective functioning.
The Reflective Function Questionnaire for Youths | 2-month
  Assesses the degree of agreement or disagreement with narratives about reflective functioning, with higher scores representing higher levels of reflective functioning.
The Reflective Function Questionnaire for Youths | 3-month
  Assesses the degree of agreement or disagreement with narratives about reflective functioning, with higher scores representing higher levels of reflective functioning.
Comfort Rating Questionnaire | Baseline
  Evaluating adverse reactions of tdcs.
Comfort Rating Questionnaire | 1-month
  Evaluating adverse reactions of tdcs.
Comfort Rating Questionnaire | 2-month
  Evaluating adverse reactions of tdcs.
Comfort Rating Questionnaire | 3-month
  Evaluating adverse reactions of tdcs.
IL-6 level | Baseline
  Detection of serum IL-6 levels using flow cytometry. The normal value is 0-5.30 pg/ml. There is a goodcorrelation between depression and elevated serum IL-6 levels.
IL-6 level | 2-month
  Detection of serum IL-6 levels using flow cytometry. The normal value is 0-5.30 pg/ml. There is a goodcorrelation between depression and elevated serum IL-6 levels.
MRI data | Baseline
  Reflecting brain structure and function
MRI data | 2-month
  Reflecting brain structure and function
EEG data | Baseline
  Reflecting brain function. It will be used for analysing Left-right asymmetry of forehead Alpha wave energy，mapping the brainnetworks.
EEG data | 2-month
  Reflecting brain function. It will be used for analysing Left-right asymmetry of forehead Alpha wave energy，mapping the brainnetworks.
TMS-evoked potentials(TEPs) | Baseline
  Reflecting cortical excitability. N15, P30, N45, P55, N100, P180 and N280 components were evoked during single-pulse TMS stimulation of motor cortex (M1). Early components of TEPs (N15-P30) reflect cortical excitatory activity, while other components (N45-N100) are associated with cortical inhibitory activity.
TMS-evoked potentials(TEPs) | 2-month
  Reflecting cortical excitability. N15, P30, N45, P55, N100, P180 and N280 components were evoked during single-pulse TMS stimulation of motor cortex (M1). Early components of TEPs (N15-P30) reflect cortical excitatory activity, while other components (N45-N100) are associated with cortical inhibitory activity.
Thinc-integrated Tools(THINC-it) | Baseline
  THINC-it（https://progress.im/en/）is the first tool to assess cognitive functioning in MDD using both subjective and objective tests and is available as a free download for use on tablets, smartphones or computers. The tool's four objective test sections use recognized cognitive paradigms to assess subjects' performance in the key cognitive domains of attention, working memory, and executive function. The Choice Reaction Time (CRT) focuses on attention and executive function, the 1-Back Memory Task (1-Back) examines memory, attention/concentration, and executive function, the Digit Symbol Substitution Test (DSST) examines processing speed, attention, and executive function, and the Test of Connectivity B (TMT-B) assesses executive function. The 5-item Cognitive Impairment Questionnaire (PDQ⁃5⁃D) is the subjective component of the instrument and can be used to assess patients' performance in attention/concentration, planning/organization, retrospection, and prospective memory.
Thinc-integrated Tools(THINC-it) | 2-month
  THINC-it（https://progress.im/en/）is the first tool to assess cognitive functioning in MDD using both subjective and objective tests and is available as a free download for use on tablets, smartphones or computers. The tool's four objective test sections use recognized cognitive paradigms to assess subjects' performance in the key cognitive domains of attention, working memory, and executive function. The Choice Reaction Time (CRT) focuses on attention and executive function, the 1-Back Memory Task (1-Back) examines memory, attention/concentration, and executive function, the Digit Symbol Substitution Test (DSST) examines processing speed, attention, and executive function, and the Test of Connectivity B (TMT-B) assesses executive function. The 5-item Cognitive Impairment Questionnaire (PDQ⁃5⁃D) is the subjective component of the instrument and can be used to assess patients' performance in attention/concentration, planning/organization, retrospection, and prospective memory.
Perceptual judgment test | Baseline
  Assess subjects' perception of interpersonal information.
Perceptual judgment test | 2-month
  Assess subjects' perception of interpersonal information.
Distance memory test | Baseline
  Assessment of Working memory.
Distance memory test | 2-month
  Assessment of Working memory.
ERP experiment | Baseline
  The participants are instructed to watch the animations，while EEG data is recorded. Event-related Mu-wave will be used for evaluating social interaction ability.
ERP experiment | 2-month
  The participants are instructed to watch the animations，while EEG data is recorded. Event-related Mu-wave will be used for evaluating social interaction ability.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China